CLINICAL TRIAL: NCT00203775
Title: Efficacy of Risperidone Versus Haloperidol in the Treatment of Aggression and Hostility in Psychotic Inmates
Brief Title: Haloperidol vs. Risperidone in the Treatment of Aggression in Psychotic Inmates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Organization: UConn Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIS-USA-269; IRB Project Number 01-250; RIS-USA-T255
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2005-05

CONDITIONS: Psychosis; Aggression
MeSH Terms: conditions — Psychotic Disorders; Aggression | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
This study examines the efficacy of haldol versus risperdal in the treatment of aggression in psychotic prison inmates. It is hypothsized that risperdal will be more effective in decreasing aggression than haldol.

ELIGIBILITY:
Inclusion Criteria:age 18 or over, psychotic disorder diagnosed on SCID, inmate at correctional facility for at least 2 weeks -

Exclusion Criteria: active withdrawal from substances of abuse, non-psychotic individuals, pregnant women, people unable to give informed consent, patients on mood stabilizers

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: catherine f lewis, md, Principal Investigator — UConn Health
Locations (1):
- University of connecticut health center, Farmington, Connecticut, United States